CLINICAL TRIAL: NCT03817281
Title: Collective Accuryn Physiologic Signals and Signatures: A Retrospective and Prospective Analysis (CAPSS Study)
Brief Title: Collective Accuryn Physiologic Signals and Signatures
Acronym: CAPSS
Status: Withdrawn | Type: Observational
Why Stopped: Lack of Enrollment
Sponsor: Potrero Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CRD-06-100473
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Critical Illness; Acute Kidney Injury; Sepsis; Septic Shock; Abdominal Compartment Syndrome
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Sepsis; Shock, Septic; Intra-Abdominal Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Accuryn Monitoring System: Observational only (no intervention). Study Cohort is patients using the Accuryn Monitoring System as a standard-of-care digital urimeter, during their standard course of treatment.
  Interventions: Device: Accuryn Monitoring System

INTERVENTIONS:
Device: Accuryn Monitoring System — The Accuryn Monitoring System is a novel Foley catheter and monitoring device capable of detecting physiologic changes in vital signs via sensors within the catheter system. These data are captured non-invasively, continuously, and at a high frequency.

SUMMARY:
The CAPSS Study is a retrospective and prospective, multi-center, single-arm post-market data collection study with an FDA cleared device. Physiologic data measurements will be collected from enrolled subjects using electronic health records and data streams via the Accuryn Monitoring System. Analysis of these data has the potential to be able to acutely guide resuscitation and monitor trends for emerging critical conditions.

DETAILED DESCRIPTION:
The primary objective of the CAPSS Study is to track and analyze changes in physiologic data streams to identify clinical signatures that may enable earlier diagnosis of, and effective intervention in, critical conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Received Accuryn Monitoring System during hospital stay.
2. Diagnosed with or developed one or more of the targeted conditions while connected to the Accuryn Monitoring System.

Exclusion Criteria:

1. In the opinion of the investigator, the patient is unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise patients from high acuity centers such as burn, trauma, surgical, and critical care units.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-29 (Actual); Primary Completion 2020-03-29 (Actual); Study Completion 2020-03-29 (Actual)

PRIMARY OUTCOMES:
Physiologic Changes | 30 days
  Track and analyze changes in physiologic data streams captured using the Accuryn Monitoring System to identify clinical signatures that may enable earlier diagnosis and effective intervention of critical conditions. Potential examples include AKI, sepsis/septic shock, ACS, and optimization of fluid resuscitation.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen M Bulger, MD, Principal Investigator — University of Washington Harborview
Locations (1):
- University of Washington Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided